CLINICAL TRIAL: NCT05216497
Title: Multicenter, Randomized, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of Ingavirin®, 90 mg Capsules in Patients With COVID-19
Brief Title: Efficacy and Safety of Ingavirin®, 90 mg Capsules in Patients With COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valenta Pharm JSC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ING-03-05-2020
Record Dates: First submitted 2022-01-28; First posted 2022-01-31 (Actual); Last update posted 2023-07-27 (Actual); Status verified 2023-07

CONDITIONS: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — pentanedioic acid imidazolyl ethanamide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ingavirin®, 90 mg capsules (Experimental): Ingavirin®, 90 mg capsules will be administered on top of standard therapy: days 1-3: 180 mg (2 capsules once a day); days 4-7: 90 mg (1 capsule 1 time per day).
  Interventions: Drug: Ingavirin®, 90 mg capsules
- Placebo (Placebo Comparator): Placebo capsules will be administered on top of standard therapy: days 1-3: 2 capsules once a day; days 4-7: 1 capsule 1 time per day.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ingavirin®, 90 mg capsules — 90-180 mg/day for 7 days on top of standard therapy
  Arms: Ingavirin®, 90 mg capsules
Drug: Placebo — 1-2 capsules for 7 days on top of standard therapy
  Arms: Placebo

SUMMARY:
The primary objective of this study is to investigate the efficacy of Ingavirin®, 90 mg capsules in achieving clinical improvement of novel coronavirus disease (COVID-19) symptoms. A secondary goal of this study is to evaluate the safety of Ingavirin®, 90 mg capsules in patients with COVID-19 infection.

ELIGIBILITY:
Inclusion Criteria:

1. Written informed consent of the patient to participate in the study.
2. Patients aged 18-75 years inclusive.
3. COVID-19 diagnosis based on laboratory confirmation of SARS-CoV-2 virus, conducted within 3 days prior to the first dose of the drug. Determination of SARS-CoV-2 virus by polymerase chain reaction (PCR) or other method regulated by the actual clinical recommendations is acceptable.
4. Patients with a mild course of COVID-19 - presence of at least 2 criteria: SpO2 ≥ 95% (mandatory criterion), body temperature ˂ 38°C, respiratory rate (RR) ≤ 22/min.
5. Duration of illness not more than 3 full days from the onset of one or more of the following symptoms until the first dose of study drug: elevated body temperature; dry cough or cough with small amount of sputum; shortness of breath; myalgia; fatigue; feeling of stuffiness in the chest; sore throat; nasal congestion/rhinorrhea; headache; feeling of heat or fever; decreased sense of smell and/or taste.
6. Presence of at least two symptoms on the COVID-19 Core Symptom Rating Scale with a score of 2 or more.
7. Women only: Negative pregnancy test result. The pregnancy test need not be performed on women who are not fertile: women who are menopausal (defined as not menstruating for at least two years or more) or who have had surgical sterilization (hysterectomy, bilateral oophorectomy, tubal ligation) or have a clinical diagnosis of infertility. The presence of surgical sterilization and infertility is evaluated on the patient's word or with a document confirming this condition.
8. Women with preserved reproductive potential and men whose partners have preserved reproductive potential agree to abstain from sexual intercourse for the duration of the study.
9. Patients who are able to understand and comply with the treatment and procedures of the study.

Exclusion Criteria:

1. Known or suspected hypersensitivity to the active ingredient or any of the excipients of the study drug.
2. Known or suspected hypersensitivity to standard therapies.
3. Presence of criteria for moderate to severe disease.
4. Need for hospitalization at the time of screening or randomization.
5. Body temperature ˂ 37.5°C.
6. Lactase deficiency, lactose intolerance, glucose-galactose malabsorption.
7. Presence of cancer within the past 2 years, or current suspicion of cancer.
8. History or current autoimmune disease.
9. Pregnancy.
10. Breastfeeding period.
11. Presence of serious lung diseases (the list can be expanded at the discretion of the investigator): moderate-to-severe bronchial asthma, severe to very severe chronic obstructive pulmonary disease (COPD), interstitial lung disease, pulmonary hypertension, pulmonary fibrosis, lung surgeries, tuberculosis (including suspected tuberculosis based on CT scan of the lungs at screening).
12. Patients with the presence of type 1 diabetes mellitus and/or decompensated type 2 diabetes mellitus.
13. Heart failure, New York Heart Association (NYHA) functional class III-IV.
14. Chronic liver failure stage II (decompensated) and higher.
15. Need for renal replacement therapy at the time of inclusion
16. History of organ transplantation.
17. History of epilepsy or need for anticonvulsant therapy.
18. Major depressive disorder, anxiety, other mental disorders requiring medication correction.
19. Acute cerebral circulation disorder, stroke, or transient ischemic attack within 90 days prior to screening.
20. Taking any antiviral and/or immunomodulatory drugs after COVID-19 manifestation.
21. Use of any immunosuppressive therapy (including tocilizumab/sarilumab) within 90 days prior to randomization, or need for immunosuppressive therapy at the time of randomization.
22. Use of anticoagulation plasma for 14 days prior to screening.
23. Use of systemic glucocorticosteroids within 90 days prior to the time of randomization, or the need to prescribe systemic glucocorticosteroids at the time of randomization.
24. History of COVID-19 vaccination.
25. Use of vaccines against viral infections within 90 days prior to the time of randomization.
26. Patients taking or having taken other experimental drugs, drugs not approved in the Russian Federation, or participating or having participated in other clinical trials within 30 days prior to screening.
27. Abuse of alcohol or psychotropic drugs and other medications currently or within the last year.
28. Patients with other serious, unstable or clinically significant medical or psychological conditions that, in the opinion of the investigator, may interfere with the patient's participation in the study.

Withdrawal Criteria:

1. Withdrawal of consent;
2. AEs that make it impossible to participate in the study or require emergency medical care in an inpatient setting (except in cases of hospitalization related to the patient's transition to a moderate to severe course of COVID-19);
3. Serious protocol violations and refusal of the participant(s) to comply with study protocol or procedures (e.g., use of protocol-prohibited therapy);
4. Pregnancy;
5. Necessity for use of medications forbidden by the protocol.
6. Participant is lost to follow-up;
7. Death of the participant;
8. Decision of the Sponsor or Investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 233 (Actual)
Dates: Start 2021-10-06 (Actual); Primary Completion 2022-01-12 (Actual); Study Completion 2022-04-25 (Actual)

PRIMARY OUTCOMES:
Time to clinical recovery | Day 2-28
  Time (in hours from first dose) to clinical recovery as assessed by Hazard Ratio analysis. Clinical recovery refers to a score of ≤1 on the COVID-19 Core Symptom Rating Scale for each symptom.

SECONDARY OUTCOMES:
Assessment of patient status | Day 2-28
  Proportion of patients with improvement of one category or more on the World Health Organization (WHO) scale by Days 2-28; proportion of patients with deterioration by one category or more on Days 2-28; average change in WHO category by Day 2-28 from baseline; proportion of patients with progression to WHO category 3 or higher by Day 14.
Assessment of clinical measures | Day 2-28
  Proportion of patients with oxygen saturation (SpO2) ≤ 93%; proportion of patients with SpO2 ˂ 95%; average change in SpO2 compared to baseline; proportion of patients with respiratory rate (RR) > 30/min; proportion of patients with RR > 22/min; proportion of patients with RR ≤ 20/min; average change in RR; proportion of patients with fever ≤ 37.0°C; proportion of patients with fever ≤ 37.5°C; proportion of patients with temperatures ≥38.5°C; mean change in temperature from baseline.
Symptom Score | Day 2-28
  Proportion of patients with a score ≤ 1 on the Daytime and Nighttime Cough Scale; average change in cough scale score from baseline; mean time to reach ≤ 1 score on the cough scale; percentage of patients with a decrease of 1 point or more on each symptom on the COVID-19 symptom scale; percentage of patients with clinical improvement (1 point or less) on each symptom on the COVID-19 symptom scale; percentage of patients with a score ≤ 1 on each symptom on the COVID-19 symptom scale; average change in score for each symptom on the COVID-19 symptom scale from baseline; average time to reach a score ≤ 1 on each symptom on the COVID-19 symptom scale.
Evaluation of laboratory and instrumental examinations | Day 2-28
  Percentage of patients negative for Severe acute respiratory syndrome-related coronavirus 2 (SARS-CoV-2) by Day 4, 8, 14, 21, 28 (if positive on previous examination); mean change in SARS-CoV-2 concentration by Day 8; time to SARS-CoV-2 elimination.

OTHER OUTCOMES:
Status assessment | Day 2-28
  Percentage of patients hospitalized during the study; length of hospitalization; proportion of patients transferred to the ICU during hospitalization; length of stay in the ICU; proportion of patients with acute respiratory distress syndrome during hospitalization; presence of fatal outcome.
Assessment of respiratory support | Day 2-28
  Percentage of patients needing oxygen therapy; percentage of patients needing high-flow oxygen therapy; percentage of patients needing noninvasive ventilation; percentage of patients needing invasive ventilation; percentage of patients needing extracorporeal membrane oxygenation (ECMO); total duration of oxygen therapy by the last day of hospitalization; total duration of high-flow oxygen therapy by the last day of hospitalization; total duration of noninvasive ventilation by the last day of hospitalization; total duration of invasive ventilation by the last day of hospitalization; cumulative duration of ECMO by the last day of hospitalization.
X-Ray evaluation | Day 2-28
  Proportion of patients with CT-1 or higher (CT-2, CT-3, and CT-4) according to lung CT data; proportion of patients with CT-0.
Safety assessment | Day 2-28
  Number and incidence of adverse events (AEs) reported during the study after study drug use and characteristics of AEs (intensity, severity, frequency, severity, expectancy, association with study therapy); number and frequency of serious adverse events (SAEs) reported during the study after the use of the study drug, and characteristics of SAEs (intensity, severity, frequency, severity, expectancy, association with the study therapy).

CONTACTS AND LOCATIONS:
Locations (14):
- Russia (14):
  - Municipal Budgetary Institution of Healthcare "Central City Hospital of Novoshakhtinsk", Novoshakhtinsk, Rostov Oblast
  - "4D Ultrasound Clinic" LLC, Pyatigorsk, Stavropol Kray
  - Ivanovo Kuvaev Clinical Hospital, Ivanovo
  - State Budgetary Institution of Healthcare of Moscow "City Polyclinic No. 2 of the Moscow Department of Healthcare", Moscow
  - Unimed-C Jsc, Moscow
  - Ryazan State Medical University named after Academician I.P. Pavlova, Ryazan
  - State Budgetary Institution of the Ryazan Region "Regional Clinical Hospital", Ryazan
  - Limited Liability Company "Medical Center "Capital-Policy", Saint Petersburg
  - Saint Petersburg State Budgetary Healthcare Institution "City polyclinic No. 112", Saint Petersburg
  - Limited Liability Company "Research Center Eco-Safety", Saint Petersburg
  - St. Petersburg State Budgetary Healthcare Institution "City Polyclinic No. 117", Saint Petersburg
  - Saint Petersburg State Budgetary Institution of Healthcare "City Pokrovskaya Hospital", Saint Petersburg
  - Astarta LLC, Saint Petersburg
  - "Family Clinic" LLC, Yekaterinburg

IPD SHARING:
Plan to Share IPD: Undecided